CLINICAL TRIAL: NCT05181228
Title: Evaluating The Effectiveness of A Family-Centered Empowerment Program Applied to Parents of Children With Oncological Problems
Brief Title: Evaluation of the Impact of a Family-Centered Empowerment Program on Self-Efficacy, Self-Esteem, Depression, Anxiety, Stress Level, and Care Skills in Parents of Children With Oncological Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Derya AKDENIZ UYSAL, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DAU_01
Record Dates: First submitted 2021-12-18; First posted 2022-01-06 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Pediatric Cancer
Keywords: Cancer; Care Ability; Family-Centered Empowerment Model; Web-Based Education; Children
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The research has a randomized controlled interventional study design. An impartial investigator who is not participating in the study will conduct the randomization. Six alternative combinations with a block size of four (ABAB(1), ABBA(2),...) containing codes A and B will be constructed using the block randomization method. From 1 to 6, combinations will be numbered. By sorting the integers (1-6) via randomizer.org 21 times in a random order, a random assignment sequence will be formed. By drawing lots with coins, it will be established which of the A and B codes is the intervention group and which is the control group. Participants who meet the inclusion criteria will be asked to sign an informed consent form, and their group will be shared with the researcher after the pre-tests (T1) are completed. In the intervention group, participants will get a web-based training based on the family-centered approach.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants were unaware of which group they were assigned to. The data will be entered using A and B codes, and the researcher doing the statistical analysis will be blind to the participants' groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Web-based family-centered empowerment program intervention) (Experimental): Intervention group participants will receive the web-based family-centered empowerment intervention for 10 weeks.
  Interventions: Behavioral: Web-Based Education Based on Family-Centered Empowerment Model
- Control Group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Web-Based Education Based on Family-Centered Empowerment Model — Parents in the intervention group will receive care for ten weeks using the family-centered empowerment model (FCEM). The first step (two weeks) is to increase knowledge. For this purpose, they will receive web-based training on cancer. The second step (four weeks) is to develop parents' self-efficacy and problem-solving skills. A web-based training and group meeting will be held to share information and experiences on the evaluation and control of the side effects of the treatment and to increase their self-efficacy in care. The third step (three week) was to increase self-esteem through participation in the training. At this stage, each participant will be asked to teach one of the family members responsible for the child's care what they have learned in the last two sessions. In the fourth step (one week), all participants in the intervention group will be evaluated by asking questions about the topics discussed in the second and third sessions and the overall content taught.
  Arms: Intervention Group (Web-based family-centered empowerment program intervention)

SUMMARY:
This study aims to develop a web-based education program based on family centered empowerment model for parents of children with oncological problems and to evaluate the effect of the program on parents' self-efficacy, self-esteem, depression, anxiety, stress level and care abilities.

DETAILED DESCRIPTION:
Cancer, one of the most important health problems of today, affects children as well as adults and the number of children diagnosed with cancer is increasing all over the world. Cancer management is generally a more complex process than other diseases and requires the caregiver family to have knowledge and skills. Because; Parents, who are the most important persons to contribute to the care of children with oncological problems, need to be supported and strengthened not only in the hospital but also in the home environment in order to manage and solve the problems and cope with this situation. One of the methods used in the empowerment of caregivers; is the family-centered empowerment model (FCEM). Model; It consists of four stages: increasing knowledge, self-efficacy and self-esteem, and evaluation. The purpose of this model; to protect the health of the family and their children, to manage the disease and symptoms, to reduce the incidence of acute attacks, to improve the quality of care by improving the quality of life of children and their parents. Because of technological advancements and growth in the number of internet users, web-based education (WBE) has become one of the most popular ways patient and family education. There is research in the literature that illustrates the benefits of web-based treatments in family strengthening.The web-based training content will be prepared based on the Family-Centered Empowerment Model. For ten weeks, parents will receive a web-based training based on the family-centered empowerment model. For the control group, routine patient education and routine hospital follow-ups will be performed by their nurses during the ten weeks follow-up period. The study's sample size; A priori power analysis was used to determine the minimum sample size. The sample size for the intervention and control groups was 38 parents, and the double-sided hypothesis was calculated as n1=n2, the effect size of 0.659, with 5% Type I error and 80% power. Research data; It was collected using the Parent and Child Information Form, the General Self-Efficacy Scale, the Rosenberg Self-Esteem Scale, the Depression Anxiety and Stress Scale, and the Care Ability Scale of Family Caregivers of Cancer Patients. A statistical package program will be used in the analysis of the data. The conformity of the mean scores of the scale to the normal distribution will be evaluated with the coefficients of kurtosis and skewness, and the means will be compared with parametric or nonparametric test techniques. The similarity of the groups in terms of demographic and clinical characteristics will be evaluated with the relevant tests. Cohen's d effect size will be calculated to express the size of the difference between the means.

ELIGIBILITY:
Inclusion Criteria:

* Being a parent (mother or father) of a child with a hematology/oncological diagnosis
* At least 1 months have passed since the child was diagnosed
* Being a parent of a child undergoing chemotherapy
* Parent who were literate
* Parents who has Internet at home
* Parents who has computer or mobile phone
* Parents who no barriers to written or verbal communication
* Parents who agree to participate in the study

Exclusion Criteria:

* Patients who do not agree to participate in the study,
* Internet not access in the home environment,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Caring Ability Of Family Caregivers Of Patients With Cancer Scale | 8 weeks
  It was developed by Nemati et al in 2020 to evaluate the care skills of caregivers involved in the care process of cancer patients and the effectiveness of empowerment interventions according to their care needs. Scale; It is a Likert-type scale consisting of 31 items, five sub-dimensions, and scored between 31 and 155. As the scale score increases, the care ability score also increases. The total scale Cronbach's alpha reliability coefficient obtained from the validity and reliability study of the scale is 0.934. The validity and reliability study of the scale in Turkey was carried out by the researcher.
General Self-Efficacy Scale | 8 weeks
  Schwarzer and Jerusalem established the General Self-Efficacy Scale in Germany in 1981. The scale's Cronbach alpha coefficient, which was adapted into Turkish in our country by Aypay (2010), was determined to be.83. The scale, which is used with people aged 12 and up, is a four-point Likert-type scale with ten items that contain statements about how well the person believes himself/herself to deal with problems in general. The score range of the scale theoretically spans between 10 and 40. If the individual achieves a high score on the scale, it suggests that his/her self-efficacy is high.
Rosenberg Self-Esteem Scale | 8 weeks
  It was developed by Morris Rosenberg in 1963 to assess self-esteem. The scale is used in adolescents, adults, and late adult individuals. In the validity and reliability study conducted by Çuhadaroğlu in Turkey in 1986, the validity coefficient was determined as 0.71. The first ten items form the self-esteem subscale and are used to evaluate self-esteem. On the scale, 0-1 points were scored as high self-esteem, 2-4 points as medium self-esteem, and 5-6 points as low self-esteem. A low score in scale scoring means high self-esteem; A high score indicates low self-esteem.
Depression Anxiety and Stress Scale | 8 weeks
  It is used to determine the depression, anxiety and stress levels of parents. Developed by Lovibond and Lovibond (1995), the first version consists of a total of 42 items. Afterwards, Henry and Crawford (2005) converted the scale into a 21-item short form. The Turkish adaptation study of the scale was conducted by Yılmaz et al. (2017) made by The scale consists of 21 items and three sub-dimensions. There are 7 questions each to measure the dimensions of depression, stress and anxiety. Each item in the scale has a 4-point scoring system that corresponds to 0, 1, 2 or 3 points according to the severity of the symptom. A minimum of 0 and a maximum of 21 points can be obtained in each dimension. High scores obtained from the sub-dimensions mean that the individual has intense feelings for the relevant sub-dimension. Cronbach's alpha internal consistency coefficients for depression, anxiety and stress sub-dimensions are .80, .81 and .75, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Yiğit, Professor, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Ciftlikkoy, Turkey (Türkiye)